CLINICAL TRIAL: NCT06421506
Title: Does Less Invasive Surfactant Administration (LISA) During High-flow Nasal Cannula Oxygen Treatment Reduces the Need for Invasive Ventilation in Late Preterm and Term Born Infants With Respiratory Distress?
Brief Title: Less Invasive Surfactant Administration in Late Preterm or Early Term Born Infants
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: King's College Hospital NHS Trust (Other)
Collaborators: Chiesi Limited (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 324607
Record Dates: First submitted 2024-05-09; First posted 2024-05-20 (Actual); Last update posted 2024-05-22 (Actual); Status verified 2024-05

CONDITIONS: Respiratory Distress Syndrome; Preterm Pregnancy; Surfactant Deficiency Syndrome Neonatal
MeSH Terms: conditions — Respiratory Distress Syndrome; Pulmonary Atelectasis

STUDY DESIGN:
Intervention Model Description: This will be a prospective single centre study with a treatment arm and a control group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Neonates given LISA during HFNC treatment (Experimental): Infants between 34-38+6 weeks gestation will receive surfactant via less invasive administration whilst on high flow nasal cannula oxygen treatment. They will have respiratory function monitoring before and after LISA.
  Interventions: Procedure: Less invasive surfactant administration during high flow nasal cannula treatment
- Neonates not given LISA (No Intervention): Infants between 34-38+6 will receive routine care and will not receive surfactant unless intubated.

INTERVENTIONS:
Procedure: Less invasive surfactant administration during high flow nasal cannula treatment — Surfactant distilled through a small tube inserted into the windpipe via the mouth whilst the baby is awake and supported with HFNC.
  Arms: Neonates given LISA during HFNC treatment

SUMMARY:
The aim of this study is to see if giving less invasive surfactant administration (LISA) during high-flow nasal cannula (HFNC) oxygen treatment reduces the need for invasive ventilation in babies with breathing problems born 2-6 weeks early.

Less invasive surfactant administration is where surfactant (a naturally produced substance which helps open up the tiny air sacs in the lungs making it easier for babies to breathe) is given into the lungs by putting a small tube into the windpipe through the mouth whilst the baby is awake. The surfactant is given slowly and breathed in.

High flow nasal cannula is a form of non-invasive support where a machine delivers warmed, moist oxygen and air through short tubes in the nose.

The investigators will be assessing whether a lower percentage of neonates need invasive ventilation within 72 hrs from birth when they have had LISA during HFNC treatment, compared to when they don't receive this treatment.

The investigators will also be looking at the length of neonatal unit stay and the cost of the stay. The investigators will also be measuring the lung function of the babies before and after they receive LISA.

DETAILED DESCRIPTION:
This study is looking at babies born 2- 6 weeks early who have breathing problems soon after birth. Some babies need to go onto a breathing machine (ventilator) or require 'non-invasive' breathing support. Either a machine delivers warmed, moist oxygen + air through short tubes in the nose (humidified high flow nasal cannula, HHFNC) or a machine delivers oxygen and air via a small mask which fits over the nose (continuous positive airway pressure, CPAP). Mechanical ventilation via a ventilator, although life-saving, can cause problems such as infection and lung injury and, therefore, whenever possible baby's breathing is supported with 'non-invasive' methods. The use of CPAP in more mature babies may also cause discomfort or lung collapse, whereas use of HHFNC may avoid those problems. The lungs of healthy full-term babies naturally produce a substance called surfactant that helps open up the tiny air sacs in the lungs and makes it easier for them to breathe. Babies born early or those with problems at birth, do not have enough of their own surfactant or it does not work properly, causing difficulty in taking in oxygen. A natural, animal-derived surfactant medication can be given into the lungs, using a small tube put into the windpipe through the mouth. This is done routinely in ventilated babies born prematurely. More recently, a technique called 'Less invasive surfactant administration (LISA)' has been developed that allows us to give surfactant to babies who are receiving 'non-invasive' breathing support (ie HHFNC) and, thus, avoiding the complications related to mechanical ventilation. A small tube is passed into the windpipe whilst the baby is awake and breathing (supported on HHFNC or CPAP) and the surfactant is slowly given and breathed into the lungs. At the moment, there have been no research studies assessing the use of LISA in more mature infants receiving HHFNC as 'non-invasive' respiratory support.

In this study the investigators want to determine if in babies born between 34 and 38+6 weeks gestation who have breathing problems and receive HHFNC oxygen treatment with LISA within 24 hours of birth will reduce the need for mechanical ventilation. The investigators will also be looking a the length on neonatal unit stay, and the cost of the stay. Lung function of the babies before and after they receive LISA will be measured.

There will be no change in the management of babies taking part in the study. Use of HHFNC, administration of LISA and respiratory monitoring is all part of routine practice. The investigators are asking for consent to analyse the routine monitoring that will be undertaken before, during and after the surfactant administration and follow up on the outcome of the baby after they have had the LISA procedure.

Surfactant is routinely used in babies and there are no extra risks from taking part in this study. HHFNC is routinely used to support babies of this gestational age who require respiratory support. There are no known or expected risks from using HHFNC with LISA but as of yet there have been no studies using this combination.

Giving surfactant may help to avoid mechanical ventilation and its side effects, but this has not been studied before in these gestational ages, hence the need for this study. Theoretically giving surfactant with HHFNC should aid even distribution of surfactant throughout the lungs whilst protecting the lungs from potential damage caused by other forms of non-invasive support such as CPAP but again there is not yet evidence supporting this.

The study will be running at King's College Hospital on the Neonatal Intensive Care Unit at the Denmark hill site and at the Local Neonatal Unit at the Princess Royal Hospital site. The study has received ethical approval and is due to commence imminently (May 2024). The study is aiming to recruit 245 patients which is estimated to take 2yrs and 4 months.

The study is funded by Chiesi Limited. The chief investigator for the study is Theodore Dassios: theodore.dassios@kcl.ac.uk

ELIGIBILITY:
Inclusion Criteria:

* Infants born at 34+0 to 38+6 weeks of gestation, requiring resuscitation at birth, but who achieve regular spontaneous breathing and have a heart rate over 100 beats per minute while receiving non-invasive support.
* Infants enrolled in the Surfon trial, born at 34+0 to 38+6 weeks of gestation, who are less than or equal to 24 hours old and exhibit signs of respiratory distress, defined as an FiO2 greater or equal to 0.30 but less than 0.45 needed to maintain an SpO2 greater than or equal to 92% or a clinically significant work of breathing regardless of the FiO2 and a clinical decision to provide non-invasive respiratory support.

Exclusion Criteria:

* Infants requiring intubation at birth
* Infants with severe congenital anomalies.

Ages: 34 Weeks to 38 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 245 (Estimated)
Dates: Start 2024-05 (Estimated); Primary Completion 2026-09 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
The percentage of neonates needing invasive ventilation within 72 hours from birth | 72 hours from birth
  The percentage of babies requiring more respiratory support and therefore needing invasive ventilation within 72 hrs from birth. The percentage from the intervention group will be compared with the control group

SECONDARY OUTCOMES:
The length of neonatal unit stay | The length of time the neonate is in hospital, up to 20 weeks
  The duration of stay on the neonatal unit will be compared between the babies receiving the intervention, and those who are not.
The cost of stay as estimated via standard NHS tariffs according to level of care | The length of time the neonate is in hospital, up to 20 weeks
  Standard NHS tariffs will be used to calculate the total cost of the stay for the babies in the intervention vs control group.
The lung function parameters two minutes before and two minutes after the administration of LISA | The first 24 hours of life
  The following lung function parameter: tidal volume will be measured for all babies receiving LISA.
The lung function parameters two minutes before and two minutes after the administration of LISA | The first 24 hours of life
  The following lung function parameter: respiratory rate will be measured for all babies receiving LISA.
The lung function parameters two minutes before and two minutes after the administration of LISA | The first 24 hours of life
  The following lung function parameter: fraction of inspired oxygen (FiO2) will be measured for all babies receiving LISA.
The lung function parameters two minutes before and two minutes after the administration of LISA | The first 24 hours of life
  The following lung function parameter: End Tidal CO2 (ETCO2) will be measured for all babies receiving LISA.
The lung function parameters two minutes before and two minutes after the administration of LISA | The first 24 hours of life
  The following lung function parameter: ratio of oxygen saturations/ fractions of inspired oxygen (SpO2/ FiO2 ratio) will be measured for all babies receiving LISA.
The SpO2/FiO2 ratio will be measured two hours after LISA administration | The first 24 hours of life
  Lung function parameter: ratio SpO2/FiO2 will be measured two hours after LISA administration for all babies receiving LISA

CONTACTS AND LOCATIONS:
Overall Officials: Theodore Dassios, PHD, Principal Investigator — King's College London

IPD SHARING:
Plan to Share IPD: No
The General Data Protection Regulation and Data Protection Act 2018 will be adhered to. Data will be anonymised before being entered into a secure database. Each participant will be issued a unique study identifier number when enrolled and this will be used on all data collection forms. Patient paper data will be stored in a locked filing cabinet in a room that is only accessible to the research team and that is based on the Neonatal Intensive Care Unit facilities at King's College Hospital. De-identified electronic patient data will be stored on encrypted computers or memory stick devices.
  On completion, the data will be analysed and a final report prepared that could be accessed via the sponsor. The study will be presented at research meetings at King's College Hospital. Anonymised study data will be presented at conferences and published by the investigators in peer reviewed journals. Participants will be notified of the outcome of the study via provision of the publication.

REFERENCES:
- [Background] Herting E, Hartel C, Gopel W. Less invasive surfactant administration (LISA): chances and limitations. Arch Dis Child Fetal Neonatal Ed. 2019 Nov;104(6):F655-F659. doi: 10.1136/archdischild-2018-316557. Epub 2019 Jul 11. PMID 31296694
- [Background] Shetty S, Egan H, Cornuaud P, Kulkarni A, Duffy D, Greenough A. Less Invasive Surfactant Administration in Very Prematurely Born Infants. AJP Rep. 2021 Jul;11(3):e119-e122. doi: 10.1055/s-0041-1735632. Epub 2021 Sep 22. PMID 34567837
- [Background] Smithhart W, Wyckoff MH, Kapadia V, Jaleel M, Kakkilaya V, Brown LS, Nelson DB, Brion LP. Delivery Room Continuous Positive Airway Pressure and Pneumothorax. Pediatrics. 2019 Sep;144(3):e20190756. doi: 10.1542/peds.2019-0756. Epub 2019 Aug 9. PMID 31399490
- [Background] Spence KL, Murphy D, Kilian C, McGonigle R, Kilani RA. High-flow nasal cannula as a device to provide continuous positive airway pressure in infants. J Perinatol. 2007 Dec;27(12):772-5. doi: 10.1038/sj.jp.7211828. Epub 2007 Aug 30. PMID 17762844
- [Derived] Jeffreys E, Jenkinson A, Kaltsogianni O, Harris C, Bhat R, Dassios T, Greenough A. Does less invasive surfactant administration during high-flow nasal cannula oxygen treatment reduce the need for invasive ventilation in late preterm and early term born infants with respiratory distress? A study protocol for a single-centre study with a treatment and control arm. BMJ Open. 2025 Jun 23;15(6):e089399. doi: 10.1136/bmjopen-2024-089399. PMID 40550714